CLINICAL TRIAL: NCT03831711
Title: A Pilot Study of 68-Ga-RM2 PET/MRI in the Evaluation of Patients With Estrogen Receptor-Positive Breast Cancer
Brief Title: 68-Ga-RM2 PET/MRI in Imaging Patients With Estrogen Receptor-Positive Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Andrei Iagaru (Other)
Collaborators: General Electric (Industry)
Responsible Party: Sponsor-Investigator, Andrei Iagaru, Professor of Radiology (Nuclear Medicine) at the Stanford University Medical Center, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-48150; NCI-2019-00237 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); BRS0098 (Other: OnCore); IRB-48150 (Other: Stanford IRB)
Record Dates: First submitted 2019-02-04; First posted 2019-02-06 (Actual); Results first posted 2023-12-13 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-11

CONDITIONS: Breast Carcinoma; Estrogen Receptor Positive
MeSH Terms: conditions — Breast Neoplasms | interventions — BAY 86-7548; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Diagnostic (68-Ga RM2, PET/MRI) (Experimental): Patients receive 68-Ga RM2 IV and after 45 minutes undergo PET/MRI over 30-60 minutes.
  Interventions: Drug: Gallium Ga 68-labeled GRPR Antagonist BAY86-7548; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Device: Investigational software and coils in PET/MR scan

INTERVENTIONS:
Drug: Gallium Ga 68-labeled GRPR Antagonist BAY86-7548 — Given IV
  Other Names: (68)-Ga-DOTA-4-amino-1-carboxymethylpiperidine-d-Phe-Gln-Trp-Ala-Val-Gly-His-Sta-Leu-NH2; 68-Ga-Bombesin Antagonist BAY86-7548; 68-Ga-DOTA RM2; 68-Ga-DOTA-Bombesin Analog BAY86-7548; [68-Ga]-labeled Bombesin Analog BAY86-7548; [68-Ga]RM2; BAY 86-7548; Ga-68-labeled Bombesin Antagonist BAY 86-7548; Gallium Ga-68-labeled GRPR Antagonist RM2
Procedure: Magnetic Resonance Imaging — Undergo PET/MRI
  Other Names: Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
Procedure: Positron Emission Tomography — Undergo PET/MRI
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging
Device: Investigational software and coils in PET/MR scan — General Electric (GE) Healthcare non-approved PET scanner coils and software

SUMMARY:
This trial studies how well 68-Ga RM2 works with PET/MRI in imaging patients with estrogen receptor-positive breast cancer. 68-Ga-RM2 is an agent used in diagnostic imaging.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the feasibility of 68-Ga RM2 PET/MRI for identification of estrogen receptor positive primary breast cancer and metastases

OUTLINE:

Patients receive 68-Ga-RM2 intravenously (IV) and after 45 minutes undergo PET/MRI over 30-60 minutes.

After completion of study, patients are followed up at 24-72 hours, and then for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* ER+ breast cancer at initial diagnosis prior to surgery or at recurrence (at least one ER+ lesion based on results of biopsy).
* Able to provide written consent
* Karnofsky performance status of ≥ 50 (or Eastern Cooperative Oncology Group (ECOG)/World Health Organization (WHO) equivalent)

Exclusion Criteria:

* Less than 18 years-old at the time of radiotracer administration
* Inability to lie still for the entire imaging time
* Inability to complete the needed investigational and standard-of-care imaging examinations due to other reasons (severe claustrophobia, radiation phobia, etc.)
* Any additional medical condition, serious intercurrent illness, or other extenuating circumstance that, in the opinion of the Investigator, may significantly interfere with study compliance
* Renal function impairment preventing administration of MRI contrast
* Metallic implants (contraindicated for MRI)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-03-19 (Actual); Primary Completion 2021-11-15 (Actual); Study Completion 2021-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrei Iagaru, Principal Investigator — Stanford Cancer Institute Palo Alto
Locations (1):
- Stanford Cancer Institute Palo Alto, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Diagnostic (68-Ga RM2, PET/MRI): Patients received 68-Ga RM2 IV and after 45 minutes undergo PET/MRI over 30-60 minutes.
Period: Overall Study
Arm/Group | Diagnostic (68-Ga RM2, PET/MRI)
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Number of lesions identified on 68Ga-RM2 PET/MRI
Arm/Group | Diagnostic (68-Ga RM2, PET/MRI)
Number analyzed (Participants) | 5
Age, Continuous [Mean (Full Range); unit: years] | 55.6 [36 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Detection of ER Positive Breast Cancer and Metastases on 68-Ga RM2 PET/MRI
Description: Number of lesions identified on 68-Ga RM2 positron emission tomography/magnetic resonance imaging (PET/MRI). The outcome will be reported as the number of participants with successful PET based detection of estrogen receptor (ER) positive breast cancer and metastases.
Time Frame: up to 2 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Diagnostic (68-Ga RM2, PET/MRI)
Number analyzed (Participants) | 5
Participants
  Breast Lesions | 4
  Lymph Node Lesions | 1

ADVERSE EVENTS:
Time Frame: up to 72 hours
Arm/Group | Diagnostic (68-Ga RM2, PET/MRI)
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

LIMITATIONS AND CAVEATS:
Early termination led to a small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-10): https://cdn.clinicaltrials.gov/large-docs/11/NCT03831711/Prot_SAP_000.pdf